CLINICAL TRIAL: NCT04687254
Title: Gender-related Characteristics of Bladder Cancer Treatment. Therapeutic Offer, Pathologic Features and Survival Outcomes of Patients Treated With Radical Cystectomy for Muscle-invasive Bladder Cancer
Brief Title: Gender-related Characteristics of Bladder Cancer Treatment
Acronym: BladderBLOG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: marco Carini (Unknown); Sergio Serni (Unknown); Andrea Minervini (Unknown); Pietro Spatafora (Unknown); Giandomenico Roviello (Unknown); Gabriella Nesi (Unknown); Ilaria Camilla Galli (Unknown); Calogero Saieva (Unknown); Graziano Vignolini (Unknown); Giovani Tasso (Unknown); Simone Morselli (Unknown)
Responsible Party: Principal Investigator, Donata Villari, Researcher, University of Florence
Other Study IDs: 18094/OSS
Record Dates: First submitted 2020-12-15; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Bladder Cancer; Radical Cystectomy; Muscle-invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most frequent cancer of the urinary tract is the bladder cancer (BC), in Italy its incidence reaches the 7% of all the new diagnosis of cancer, accounting for the fifth cause of death in the western countries, overall 140.000 new cases per year in Europe. In the year 2017, the Italian association for medical oncology (AIOM) recorded in our country about 21.700 new diagnosis of BC men and 5.300 in women. This data show not only a relevant gender disparity on the disease incidence (in 5th to 7th decade male incidence: 11-12% of all new diagnosis of cancer versus 1% in women) but also on the outcomes of treatment. Overall, the 30% of all the new diagnosis have a muscle-invasive (MIBC) onset, the female gender suffer a correlation with a more advanced disease at the time of first diagnosis. As a consequence, men have lower BC-related mortality when compared to women (p<0,001). This discrepancy in the mortality rate has been investigated by many authors, resulting in the evidence that female gender suffers higher risks, especially during the first two-years after the radical cystectomy. A comprehensive explanation has not been formulated yet, but a multiplicity of cofactors, including variations in the hormone receptors and tumor biology as well as the different anatomy between male and female, have been identified as potentially relevant. Another important issue in the pre-operatory management of female patients with BC is the misleading interpretation of hematuria. It seems to directly correlate with the evidence that women suffer a more advanced stage at diagnosis, and this element has been withheld in the list of relevant risk factors for prognosis. Nevertheless, a thorough analysis of their effect will only be possible in the future, as well-designed prospective and randomized clinical trials are currently not available.

A part from the preoperatory disparity, it has also been described that men are more frequently candidates to an orthotopic urinary diversion, leading female patients to an irreversibly altered perception of personal integrity and body image, namely to a lower quality of life after radical cystectomy. The female anatomy has been considered as a limitation to continence recovery, resulting in preoperative counselling more frequently against in favor of ileal conduit or not-continent urinary diversions.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing radical cystectomy since September 2016 December 2020
* Development of bladder cancer confirmed histologically
* Written informed consent

Exclusion Criteria:

• Lack of clinical and prognostic data on selected patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with radical cystectomy for muscle-invasive bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
gender-related discrepancies in the treatment offer for patients affected by MIBC from September 2016 to December 2020 | 36 months

SECONDARY OUTCOMES:
gender-related difference in the clinical and pathologic features of MIBC | 36 months
gender-related difference in the survival outcomes | 36 months
gender-related difference in the risk factors for development of BC | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Donata Villari, Florence, FI, Italy